CLINICAL TRIAL: NCT02651194
Title: A Single-Arm, Open-Label, Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Renally-Impaired Adults With Chronic Hepatitis C Virus Genotype 1 - 6 Infection (EXPEDITION-4)
Brief Title: A Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Renally Impaired Adults With Chronic Hepatitis C Virus Genotype 1 - 6 Infection
Acronym: EXPEDITION-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-462; 2015-002353-35 (EudraCT Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Chronic Hepatitis C Virus (HCV) Infection
Keywords: Treatment-naïve; HCV Gentoype 2; Non-cirrhotic; Chronic Hepatitis C; HCV Gentoype 5; HCV Gentoype 4; HCV Gentoype 6; HCV Gentoype 1; Compensated cirrhotic; Treatment-experienced; HCV Gentoype 3
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-493/ABT-530 (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 12 weeks of treatment with the ABT-493/ABT-530 combination regimen in adults with chronic HCV genotype 1 - 6 infection and chronic severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV) infection
* Screening laboratory results indicating HCV genotype 1 - 6 (GT1 - 6) infection.
* Subject must be HCV treatment-naïve or have failed previous HCV treatment.
* Subjects with underlying chronic renal impairment (estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 as estimated by the MDRD method at screening, including those requiring dialysis).
* Non-cirrhotic subjects must have documented absence of cirrhosis and subjects with cirrhosis must have documented compensated cirrhosis.

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any excipients of the study drug.
* Female who is pregnant, planning to become pregnant during the study, or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
* HCV genotype performed during screening indicating co-infection with more than 1 HCV genotype; HCV GT3 infected, treatment-experienced subjects were excluded.
* Patients who failed a previous regimen containing protease inhibitor (PIs) and/or nonstructural protein 5A (NS5A) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- [Derived] Gane E, Lawitz E, Pugatch D, Papatheodoridis G, Brau N, Brown A, Pol S, Leroy V, Persico M, Moreno C, Colombo M, Yoshida EM, Nelson DR, Collins C, Lei Y, Kosloski M, Mensa FJ. Glecaprevir and Pibrentasvir in Patients with HCV and Severe Renal Impairment. N Engl J Med. 2017 Oct 12;377(15):1448-1455. doi: 10.1056/NEJMoa1704053. PMID 29020583
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 35-day screening period.
Period: Overall Study
Arm/Group | ABT-493/ABT-530
Started | 104
Completed | 99
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug (ITT population).
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.52 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 104
percentage of participants | 98.1 [95.4 to 100.0]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: up to 12 weeks
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 104
percentage of participants | 0.0 [0.0 to 3.6]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 100
percentage of participants | 0.0 [0.0 to 3.7]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ABT-493/ABT-530
Serious Adverse Events (participants affected / at risk) | 25/104
Other Adverse Events (participants affected / at risk) | 54/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 (N=104)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3
HYPERTENSIVE CARDIOMYOPATHY (Cardiac disorders) | 1
MITRAL VALVE STENOSIS (Cardiac disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1
CATHETER SITE INFECTION (Infections and infestations) | 1
ERYSIPELAS (Infections and infestations) | 1
INFECTED FISTULA (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
RENAL ABSCESS (Infections and infestations) | 1
WOUND INFECTION (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1
FACIAL PARESIS (Nervous system disorders) | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1
END STAGE RENAL DISEASE (Renal and urinary disorders) | 1
RENAL HAEMORRHAGE (Renal and urinary disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
HAEMATOMA (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 2
SUPERIOR VENA CAVA OCCLUSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 (N=104)
DIARRHOEA (Gastrointestinal disorders) | 10
NAUSEA (Gastrointestinal disorders) | 11
VOMITING (Gastrointestinal disorders) | 8
ASTHENIA (General disorders) | 10
FATIGUE (General disorders) | 15
DECREASED APPETITE (Metabolism and nutrition disorders) | 9
DIZZINESS (Nervous system disorders) | 7
HEADACHE (Nervous system disorders) | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.